CLINICAL TRIAL: NCT01385813
Title: Inflammatory Markers in Preeclampsia
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Professor Lars Mørkrid, University of Oslo
Other Study IDs: INFLAMMARPE11
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-05

CONDITIONS: Preeclampsia
Keywords: pre-eclampsia; inflammatory markers; serological biobank; To assess whether the inflammatory markers could be useful; in order to identify pregnant women at risk to; develop preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women who develop preeclampsia: pregnant women who develop preeclampsia (n =43) compared to pregnant women fulfilling a normotensive pregnancy (n= 86).

SUMMARY:
This is an investigation of inflammatory markers in women destined to develop preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian origin

Exclusion Criteria:

* Previous diseases e.g. cardiovascular disease, diabetes, hypertension, inflammatory bowel disease, serious organ disease

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study comprised 43 pregnant women who developed preeclampsia and 86 pregnant women who fulfilled a normotensive pregnancy.
  All women were of Caucasian origin, and were nulliparous.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 1999-01; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)